CLINICAL TRIAL: NCT00882037
Title: Risk and Protective Factors for Rural Methamphetamine Dependence
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0335-08-FB
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine Dependence; Substance Abuse Treatment; Rural and Urban; Latino and Non-Latino

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meth Dependence: Methamphetamine Dependence in residential Substance Abuse Treatment Program

SUMMARY:
The primary goal of this study is to identify factors which may put a person that has used methamphetamine at greater risk for mental and physical health problems and social problems and factors that may lessen the risk for these problems. This study will also compare methamphetamine use between Latino and non-Latino persons and those that live in a rural area or urban area. The investigators hypothesis is that rural persons with methamphetamine dependence will have greater socio-demographic, bio-psychosocial and behavioral risk factors than their urban counterparts.

DETAILED DESCRIPTION:
Methamphetamine (meth) is second only to alcohol as the primary drug of abuse in persons entering substance use disorders (SUD) treatment in rural Nebraska 1 . The National Survey on Drug Use and Health 2002-2005 (NSDUH) found meth use increased as the setting became more rural 2 . In a previous study comparing rural and urban persons with meth use disorders (MUD), we found significant differences, with rural persons reporting earlier first regular use of meth, greater meth-related psychotic symptoms, more alcoholism, and more intravenous (IV) use 3 . No studies have compared frequency of other behavioral risk factors in rural and urban meth users. Similarly, no studies have compared risk factors for methamphetamine dependence in this uniquely rural drug use disorder. It is critical that other high risk behaviors (in addition to IV use) be identified in rural persons with MUD and that risk factors for MUD be identified as a crucial first step in providing resources to tailor prevention efforts in rural populations.

In addition to the need for further research on risk factors, scholars have called for more studies on protective factors to develop more effective intervention programs 4 . Researchers have identified factors that mitigate negative outcomes among individuals at high risk. In general, active coping and high levels of social support and empathy have been linked to better health outcomes whereas avoidance coping and low levels of social support and empathy have been associated with worse health outcomes 4, 5 . However, no factors have been identified in rural meth users which are protective for worse health outcomes.

Meth distribution has been linked to "Mexican Drug Trafficking Organizations" and "Hispanic polydrug trafficking organizations" 6, 7 , but there is little research examining meth use in Latinos. In a previous study of Hispanic and non-Hispanic white individuals with MUD, Hispanics reported less education and more employment problems, 8 but the study did not address rural MUD. This proposed study of rural and urban Latinos with meth dependence will provide initial data to begin to inform prevention efforts targeting rural Latinos with MUD and may be useful in rural Latinos with other SUD.

Our interdisciplinary investigative team proposes to address the following Specific Aims over a two-year period: 1) compare socio-demographic, bio-psychosocial and behavioral risk and protective factors between rural and urban persons with methamphetamine dependence (Year One); 2) identify factors that place persons with methamphetamine dependence at risk for greater psychopathology and identify factors that mitigate those persons from psychopathology (Year One); 3) compare severity of methamphetamine dependence between Latino and non-Latino populations and urban and rural Latino populations (Year Two). Our hypothesis is that rural persons with methamphetamine dependence will have greater socio-demographic, bio-psychosocial and behavioral risk factors than their urban counterparts.

The targeted populations will be adults with methamphetamine dependence. We will enroll 150 individuals (75 rural and 75 urban) 75 of whom will be Latinos from substance abuse treatment sites. Data analyses will focus on comparing MUD across urban/rural and Latinos/non-Latinos. Thus, this study will identify factors which may place rural, urban, Latino, and non-Latino persons with MUD at greater risk for, or protect them from, psychopathology, infectious complications, and poorer treatment outcome. The long-term goals of this study are to: a) provide data that will strengthen a re-submission to the National Institute on Drug Abuse (Behavioral and Social Science Research on Understanding and Reducing Health Disparities, PAR-07-379 ); b) establish relationships with providers of substance abuse treatment to Latinos facilitating enrollment of Latinos in future research studies; and c) identify specific factors that can be incorporated into prevention strategies in underserved populations (e.g. Latinos, rural populations).

ELIGIBILITY:
Inclusion Criteria:

* Adults in SUD treatment facilities meeting DSM-IV criteria for methamphetamine dependence and able to provide informed consent.
* We intend to oversample Latinos in order to achieve a group with sufficient power to compare to non-Latinos. Our goal is to recruit 75 Latinos and 75 non-Latinos.

Exclusion Criteria:

* Persons not meeting the DSM-IV criteria for methamphetamine dependence and persons unable to complete informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a study of 150 rural and urban persons in treatment for methamphetamine dependence. We propose to enroll 150 participants (75 rural and 75 urban) over a two year period. Of these 150 participants, 75 will be Latino and 75 non-Latino (approximately 37 rural and 37 urban for each group).
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-12-12 (Actual); Primary Completion 2010-12-15 (Actual); Study Completion 2010-12-15 (Actual)

PRIMARY OUTCOMES:
Rural v urban persons with methamphetamine dependence entering SUD treatment | Year 1
  Compare socio-demographic, bio-psychosocial and behavioral risk and protective factors between rural and urban persons with methamphetamine dependence entering SUD treatment.

SECONDARY OUTCOMES:
Latino v non-Latino persons with methamphetamine dependence | Year 2
  Compare methamphetamine dependence between Latino and non-Latino populations and examine methamphetamine dependence among urban and rural Latino populations.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Grant, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Saint Francis Medical Center Alcohol and Drug Treatment Center, Grand Island, Nebraska
  - Catholic Charities - Campus for Hope, Omaha, Nebraska